CLINICAL TRIAL: NCT04899648
Title: Hypertension Prevention Program, Implementation and Scale up- a Hybrid Effectiveness Implementation Study in Schools of Dhulikhel and Banepa
Brief Title: Hypertension Prevention Program, Implementation and Scale up- a Hybrid Effectiveness Implementation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Bhawana Shrestha, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00012777
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Hypertension; Dietary Modification; Health Behavior
Keywords: Hypertension Prevention
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Experimental): Receives nutrition and exercise intervention classes
  Interventions: Behavioral: Behavioral Intervention Group
- Control Group (No Intervention): Does not receive any intervention classes

INTERVENTIONS:
Behavioral: Behavioral Intervention Group — Behavioral intervention: (a) form groups and choose peer leaders; (b) train peer leaders on 16 core classes based on diabetes prevention program curriculum; (c) support and motivate peer leaders to lead intervention in their group; (d) monitoring of the interventions.
  Arms: Behavioral Intervention

SUMMARY:
This is an effectiveness-implementation study to assess the effectiveness of a peer-led multi-component lifestyle program that will aim to lower BP among pre-hypertensive individuals in Nepal. The program will aim to encourage weight loss, improve diet (using a DASH diet), lower sodium intake, encourage only moderate alcohol intake among drinkers, and encourage more physical activity through peers.

DETAILED DESCRIPTION:
Hypertension is a serious medical condition and can increase the risk of heart, brain, kidney and other diseases. It is a major cause of premature death worldwide, with upwards of 1 in 4 men and 1 in 5 women - over a billion people - having the condition. The burden of hypertension is felt disproportionately in low- and middle-income countries, where two-thirds of cases are found, largely due to increased risk factors in those populations in recent decades Pre-hypertension, defined as systolic blood pressure (BP) of 120-139 mmHg or diastolic BP of 80-89 mmHg, is a precursor to hypertension, and is associated with excess morbidity and deaths from cardiovascular diseases (CVD). Hence, the reduction of BP to optimal levels is a major public health priority. Although clinical trials have shown that pharmacotherapy lowers BP among pre-hypertensives; it has been argued that pharmacotherapy is not reasonable because the absolute risk in patients without other CVD risk factors is low and pharmacotherapy is costly. Lifestyle modifications have proven to reduce BP, and are also useful to prevent other chronic diseases. Major lifestyle modifications shown to lower BP include weight loss; reduced sodium intake; regular aerobic physical activity; moderate alcohol drinking; the Dietary Approach to Stop Hypertension diet - a diet rich in fruits, vegetables, low-fat dairy products, potassium and calcium, and reduced dietary cholesterol, saturated and total fats. Combinations of two or more lifestyle modifications may have even better results. However, most of the studies have focused on one or two lifestyle interventions and are tested in efficacy trials in a clinical setting. Therefore, there is a major gap in the evidence for the effectiveness of a community-based multi-component intervention on BP reduction. In addition, it is not clear how such an intervention would be scaled up to the general population in low-and-middle-income countries, where the burden of hypertension and CVD is the highest.

To address this gap, the investigators propose to conduct an effectiveness-implementation study to assess the effectiveness of a peer-led multi-component lifestyle program that will aim to lower BP among pre-hypertensive individuals in Nepal. The program will aim to encourage weight loss, improve diet (using a DASH diet), lower sodium intake, encourage only moderate alcohol intake among drinkers, and encourage more physical activity through peers. Peer education can be as effective as using health professionals and is a cost-effective and sustainable method for lifestyle modification. The peer-education approach is driven by social learning theory, emphasizing credibility, role modeling, empowerment, and reinforcement which contrasts with the delivery of lifestyle modification advice in the usual clinical setting. While implementing the peer-led multi-component lifestyle intervention, the investigators will collect information on factors affecting the delivery of the program and the potential for scaled-up implementation in a real-world situation. The feasibility and scalability of such programs in a real-life setting have not been studied. Besides, there are three key challenges to manage pre-hypertension and hypertension in low-and middle-income countries (LMICs). First, the pre-hypertensive population is considered non-diseased; hence they are not in contact with the health system. Second, even though the efficacy of lifestyle modifications has been proven, sustainable lifestyle modifications in the general population are difficult to achieve due to the complexity of behavioral change. And third, the health system in LMICs is already worn out due to the double burden of disease, and inadequate financing and human resources. To address this massive challenge in an LMIC such as Nepal, a cost-effective, community-based, sustainable, and scalable intervention is required. The proposed study will establish evidence for a new model to lower BP in a community setting, by determining the effectiveness of the peer-led multi-component program and informing the success of implementation and scalability. This model will provide a valuable resource for making recommendations and dissemination plans to implement and sustain lifestyle interventions for lowering BP at the community level.

As such, the objectives of this study are:

1. To measure the effectiveness of the peer-led online multi-component lifestyle program on reducing BP among the school employees of Dhulikhel and Banepa, Nepal. The investigators will compare the change in systolic BP at twelve months between the peer-led multi-component program group and usual care group using a community-based cluster randomized control trial.
2. To measure the success of implementation and inform the scalability of the peer-led multi-component lifestyle program. The investigators will evaluate (a) program adoption by assessing changes in weight, diet, and physical activity behaviors among lifestyle intervention participants; (b) fidelity to the program design by assessing activities of peer-educators; and (c) acceptability of the program through (i) in-depth, semi-structured interviews with lifestyle intervention program dropouts; and (ii) focus group discussions with lifestyle intervention program participants.
3. To assess the impact of Covid-19 in hypertension management in context to the mental wellbeing of hypertensive patients. The investigators will measure the impact of Covid-19 on the mental health of a participant by measuring their anxiety and depression levels through a questionnaire scale.

After identification of possible participants, the principal investigator and/or the research assistants would make formal phone calls to the principals of the different educational institutes to describe the research project. The principals of the educational institutes are, then, sent information sheets and other informational materials regarding the project via email. Then, after the approval of the principal, all the staff of the educational institutions would be sent an information sheet and other information regarding the project. After everyone is informed, a formal zoom or google meet appointment would be made with all the staff of the educational institute. In this manner, the study participants would be recruited and screened.

After 500 participants are selected from various educational institutes, their baseline information will be collected which would include aspects of their demography, physical activity, behavioral history like smoking and alcohol consumption, diet recall, mental health status and anthropometric measurements. This will all take place in the first 3 months of the study. All of this information will be collected via an online survey. As for the anthropometric measurements, the investigators will have provided anthropometric instruments like Digital Blood Pressure Machine, Digital Weighing Scale and Mechanical Measuring tape, to each educational institute and also provided them with World Health Organization Guidelines to use those instruments. Using the tools provided by the investigators, the study participants will measure their anthropometric data themselves when they are in their workplace. This information is then sent along with their other information while filling up the online survey. After that, a computer-generated randomization process will be carried out after which 250 participants will be selected for the intervention process.

Control Group: The remaining 250 Participants in the control group would not get exercise and nutritional classes. But they will all get the study and educational material regarding hypertension prevention after the end of the study.

Behavioral Classes: Participants (n=250) who are selected for the Behavioral Intervention classes will be connected with the study team for 20 minutes video, 20 minutes of discussion and 20 minutes of exercise every week. It would include 16 core sessions weekly during the next four months of the program followed by 1 month maintenance sessions. Each core session will last 1 hour every week. The audio and video of the sessions for some intervention groups will be recorded. These Participants would also be reimbursed Nrs. 50 for the data package 16 times.

Peer Leader: Among the selected participants from the Intervention group, 10% of the participants would be appointed peer leaders. The peer leaders will go through health education classes via online platforms using various videos and presentations. The peer leaders will also be paired with the professional health educators from the study staff and will be informed about aspects like Diabetes Prevention Program Curriculum along with dieting and exercise classes. Professional health educators will train the peer educators and provide online supervision as well. The health educators will also assess the classes taken by peer leaders to the rest of the participants and provide necessary feedback and motivation. Behavior intervention will be comprised of extensive education sessions, group counseling and goal setting and monitoring exercises based on the diabetes prevention program developed by India Works. Peer Leader will conduct 16 session classes for the remaining participants in the intervention group virtually. Peer Leader will measure Blood Pressure, Height and weight of the Participants once a month from the Intervention Group.

Endline: This survey will be done for all the participants both in the control and intervention groups. This would take 15-20 minutes. Some of the questions from the baseline survey will be filled by the participants. (about daily activities, cigarettes and alcohol intake) Height, weight, blood pressure will be accessed by themselves or their designated peer leader. Questions about 24 hours diet, physical activities will be asked by the research assistants through online platforms like zoom or viber.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employees who work a minimum of 40 hours per week as appointed by the school within the age group of 18-60 including both male and female.

Exclusion Criteria:

* Pregnant females, Participants below 18 years or and above 60.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-05-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood pressure | Four months
  An average of three measurements, mmHg continuous variable
Diastolic Blood pressure | Four months
  An average of three measurements, mmHg continuous variable

SECONDARY OUTCOMES:
Body Mass Index | Four Months
  Change in Weight to Height ratio based on BMI
Healthy food intake | Four Months
  Intake of whole grains, fruits and vegetables based on 24 hour diet recall

CONTACTS AND LOCATIONS:
Overall Officials: Bhawana Shrestha, MPH, PhD, Principal Investigator — University of Washington